CLINICAL TRIAL: NCT05455008
Title: Feasibility, Acceptability, and Preliminary Efficacy of a Single-arm, Remotely-delivered Health Coaching Intervention to Increase Physical Activity and Reduce Sedentary Behavior During Pregnancy
Brief Title: INcreasing Steps in PREgnancy Study
Acronym: INSPiRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Iowa Fraternal Order of Eagles (Unknown)
Responsible Party: Principal Investigator, Kara Whitaker, Assistant Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201910845
Record Dates: First submitted 2022-06-27; First posted 2022-07-13 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Pregnancy Related; Exercise; Sedentary Behavior; Behavior and Behavior Mechanisms
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Behavior

STUDY DESIGN:
Intervention Model Description: Single-arm remotely-delivered health coaching pilot intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remotely-delivered health coaching intervention (Experimental): Single-arm remotely-delivered health coaching intervention to increase physical activity and reduce sedentary behavior during pregnancy, consisting of 12 health coaching sessions.
  Interventions: Behavioral: Remotely-delivered health coaching intervention

INTERVENTIONS:
Behavioral: Remotely-delivered health coaching intervention — Single-arm remotely-delivered health coaching intervention to increase physical activity and reduce sedentary behavior during pregnancy, consisting of 12 health coaching sessions.

SUMMARY:
This pilot study will test the feasibility, acceptability, and efficacy of a remotely-delivered intervention for increasing daily physical activity levels and reducing sedentary behavior during pregnancy among women who are insufficiently active (i.e. reporting <150 minutes/week of moderate intensity activity and/or <7,000 steps/day). It is hypothesized that women will increase daily steps and decrease total sedentary time across the second trimester of pregnancy.

DETAILED DESCRIPTION:
Physical activity during pregnancy is safe for the mother and baby and has many health benefits; however, less than 25% of pregnant women meet the recommended physical activity guidelines. Data from the investigative team also indicates that high sedentary behavior across pregnancy trimesters is associated with an increased risk of hypertensive disorders of pregnancy and other adverse pregnancy outcomes, independent of physical activity level. There is a clear need to encourage physical activity participation while concurrently promoting a reduction in sedentary time during pregnancy.

This pilot study will test the feasibility, acceptability, and efficacy of a remotely-delivered intervention for increasing daily physical activity levels and reducing sedentary behavior during pregnancy among women who are insufficiently active (i.e. reporting <150 minutes/week of moderate intensity activity and/or <7,000 steps/day). We hypothesized that participants would increase daily steps and decrease total sedentary time over the course of the intensive intervention phase (second trimester, ~14 weeks). Further, we hypothesized that participants would maintain or have minimal changes in daily steps and total sedentary time from the end of the intensive intervention phase through the follow-up phase (third trimester, ~14 weeks).

Intervention Summary: Participants have 12 contacts with a health coach using a telehealth platform to provide ongoing support and discuss physical activity and sedentary behavior goals based on real-time data obtained from a Fitbit monitor. Intervention contacts will be weekly for the first month, bi-monthly in months 2-4, and monthly until delivery. Participants will also receive one text message between each intervention contact to reinforce content discussed in coaching sessions. Physical activity and sedentary time will be assessed objectively using an activPAL device for 7-days at baseline and at the end of the intensive intervention phase (second trimester, ~14 weeks).

Specific Aims:

Aim 1: To test the feasibility of a remotely-delivered intervention designed to increase physical activity levels and reduce sedentary behavior during pregnancy. Feasibility will be defined by: (1) recruitment and enrollment of at least 50% of eligible women who completed the screening form, (2) retention of 85% or more participants from baseline through delivery, (3) adherence if participants attended 75% or more of the health coaching sessions on average and wore and synced their Fitbit device on at least 75% of days from baseline through the end of the intervention.

Aim 2: To test the acceptability of a remotely-delivered intervention designed to increase physical activity levels and reduce sedentary behavior during pregnancy. Acceptability will be defined as at least 75% of the participants indicating they were satisfied or very satisfied with the program overall.

Aim 3: To test the preliminary efficacy of a remotely-delivered intervention designed to increase physical activity levels and reduce sedentary behavior during pregnancy. Efficacy will be determined using paired t-tests to assess activPAL-measured changes in physical activity (steps/day, stepping minutes/day, standing minutes/day) and sedentary behavior (sedentary minutes/day, total and in bouts of 30 and 60 minutes) from baseline through the end of the second trimester (intensive intervention phase). The intervention specifically aims to increase physical activity levels and reduce sedentary behavior from enrollment through the end of the second trimester of pregnancy (intensive intervention phase), and then will encourage participants to maintain activity levels based on their comfort level through the third trimester (follow-up phase).

ELIGIBILITY:
Inclusion Criteria:

* less than 13 weeks pregnant
* between 18-44 years of age
* owned smart phone
* able to speak, comprehend, read, and write in English
* self-reported insufficient activity as determined by the PARmed-X for pregnancy (exercising less than 150 minutes per week) and less than 7,000 steps/day

Exclusion Criteria:

* currently enrolled in another research study about exercise
* physical limitations that prevented exercise
* instructed by a physician to not exercise during pregnancy
* hospitalized for a psychiatric disorder in the past six months
* absolute or relative contraindication to exercise as determined by the PARmed-X for pregnancy
* other serious medical conditions
* averaged <9,000 steps/day as determined by the activPAL device worn prior to the first coaching session

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility: recruitment and enrollment | Through study completion, an average of 28 weeks
  Feasibility will be defined by recruitment and enrollment of at least 50% of eligible women who completed the screening form
Feasibility: retention | Through study completion, an average of 28 weeks
  Feasibility will be defined by retention of 85% or more participants from baseline through delivery
Feasibility: adherence | Through study completion, an average of 28 weeks
  Feasibility will be defined by adherence if participants attended 75% or more of the health coaching sessions on average and wore and synced their Fitbit device on at least 75% of days from baseline through the end of the intervention.
Acceptability | Through study completion, an average of 28 weeks
  Acceptability will be defined as at least 75% of the participants indicating they were satisfied or very satisfied with the program overall.
Efficacy - changes in physical activity (steps/day) | Across the second trimester (intensive intervention phase), an average of 14 weeks
  Preliminary efficacy will be determined using paired t-tests to assess activPAL-measured changes in physical activity (steps/day).
Efficacy - changes in sedentary time (min/day) | Across the second trimester (intensive intervention phase), an average of 14 weeks
  Preliminary efficacy will be determined using paired t-tests to assess activPAL-measured changes in sedentary behavior (sedentary minutes/day).

SECONDARY OUTCOMES:
Efficacy - changes in physical activity (stepping min/day and standing min/day) | Across the second trimester (intensive intervention phase), an average of 14 weeks
  Preliminary efficacy will be determined using paired t-tests to assess activPAL-measured changes in physical activity (stepping minutes/day, standing minutes/day)
Efficacy - changes in sedentary time (sedentary min/day in bouts of 30 and 60 minutes) | Across the second trimester (intensive intervention phase), an average of 14 weeks
  Preliminary efficacy will be determined using paired t-tests to assess activPAL-measured changes in sedentary behavior (sedentary minutes/day in bouts of 30 and 60 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through the University of Iowa data repository
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available after publication of the primary outcomes
Access Criteria: Open access to de-identified data.
URL: https://iro.uiowa.edu/esploro/outputs/dataset/9984236057502771

REFERENCES:
- [Background] Whitaker KM, Jones MA, Dziewior J, Anderson M, Anderson C, Gibbs BB, Carr LJ. Feasibility, acceptability, and preliminary efficacy of a single-arm, remotely-delivered health coaching intervention to increase physical activity and reduce sedentary behavior during pregnancy. BMC Pregnancy Childbirth. 2022 Oct 2;22(1):740. doi: 10.1186/s12884-022-05073-4. PMID 36184599
- Available data/document: Individual Participant Data Set — https://iro.uiowa.edu/esploro/outputs/dataset/9984236057502771